CLINICAL TRIAL: NCT06741137
Title: A Pilot Study of the Effect of the Combination of Inhaled Nitric Oxide and Prone Position Under EIT Monitoring on Efficacy in Patients with ARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024ky074
Record Dates: First submitted 2024-12-16; First posted 2024-12-18 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-10

CONDITIONS: ARDS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- inhaled nitric oxide combined with prone position ventilation (Experimental)
  Interventions: Procedure: inhaled nitric oxide combined with prone position ventilation

INTERVENTIONS:
Procedure: inhaled nitric oxide combined with prone position ventilation — inhaled nitric oxide combined with prone position ventilation

SUMMARY:
Investigating the Impact of Combined Inhaled Nitric Oxide and Prone Positioning on the Efficacy in ARDS Patients

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years;
2. Patients with moderate to severe ARDS on mechanical ventilation

Exclusion Criteria:

1. Patients with severe asthma or acute exacerbation of chronic obstructive pulmonary disease (COPD), lung tumors, post-lung resection, and post-lung transplantation.
2. Patients with hemodynamic instability requiring vasopressor support: dopamine or dobutamine >15 µg/kg/min, norepinephrine >0.3 µg/kg/min.
3. Cardiogenic pulmonary edema.
4. Patients with severe facial deformities, facial trauma, or severe thoracoabdominal trauma that precludes prone positioning ventilation.
5. Mid to late pregnancy.
6. Patients with a history of malignancy or other irreversible diseases/conditions, including those in the terminal stage.
7. Patients expected to be discharged soon or requiring invasive mechanical ventilation for less than 24 hours.
8. Patients currently participating in other studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intratidal gas distribution | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China